CLINICAL TRIAL: NCT00583960
Title: Office-based Radial Expansion Balloon Dilation of the Esophagus and Trachea
Status: Withdrawn | Type: Observational
Why Stopped: PI chose not to proceed with study.
Sponsor: University of California, Davis (Other)
Responsible Party: Peter Belafsky, MD, Ph.D., University of California Davis
Other Study IDs: 200715177-1
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Tracheal Stenosis
Keywords: swallowing problems; tracheal stenosis
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective chart review of UCDMC patients who have undergone esophageal or tracheal balloon dilation to record data including age, gender, diagnosis pre-and post-procedure eating assessment tool, esophagoscopy findings, tracheobronchoscopy findings, and pre-and post-procedure videofluoroscopic findings.

DETAILED DESCRIPTION:
Dilation of the esophagus is performed for strictures, webs, and rings at all levels of the esophagus. Dilation of the trachea is performed for subglottic and tracheal stenosis. Radial expansion balloons have been developed by Bost Scientific Corporation for the purpose of dilating the esophagus and trachea through flexible esophagoscopies. These sequential controlled radial-expansion balloons can be introduced via a guide wire through the working channel of a 5.1 mm transnasal esophagoscope. Traditionally, otolaryngologists have performed esophageal and tracheal dilation per oral under general anesthesia. This technique allows the procedure to be performed in the office, sparing the patient the risk of anesthetics. The purpose of this study is to review the UCDMC experience with esophageal and tracheal balloon dilation using the transnasal esophagoscope.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone esophageal or tracheal balloon dilation since 1/1/05
* patients who underwent an attempted dilation since 1/1/05

Exclusion Criteria:

* Younger than 18 years of age
* Those who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UCDMC Otolaryngology Voice and Swallowing Center patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD, PhD, Principal Investigator — University of California, Davis